CLINICAL TRIAL: NCT01042431
Title: Nutrition Day in Hospitals, Nursing Homes and Community. Israel January 2010
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Y. Folman, Director Orthopedic B' Ward, Hillel Yaffe Medical Center
Other Study IDs: 0057-09-HYMC
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Nutritional Status
Keywords: Nutritional status of ward patients and hospitalization outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ward population: Patients hospitalized in the Orthopedics B Ward in the Hillel Yaffe Medical Center that choose to participate in the study
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
This study is a one-day international cross-sectional nutritional audit in one ward. The purpose of this study is to generate a risk and level of nutritional intervention profile for an individual unit/ward based on case-mix, structures and social environment.

ELIGIBILITY:
Inclusion Criteria:

* A adult patients within the unit from 7H00 to 7H00

Exclusion Criteria:

* Patients younger than 18 years
* Patients admitted and discharged during same calendar day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Orthopedic B' Ward
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel